CLINICAL TRIAL: NCT02029079
Title: The Effect of Food and Beverage Based Nutritional Supplements in Recipients of Home Care Services at Risk of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013/962
Record Dates: First submitted 2013-12-18; First posted 2014-01-07 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2014-01

CONDITIONS: Malnutrition
Keywords: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E+ drink, enriched with energy and nutrients. (Experimental): The intervention consists of 300 ml E+ per day for 35 days in addition to a normal food intake. This means 525 kcal, and 22.5 gram protein extra per day for five weeks.
  Interventions: Dietary Supplement: E+
- Control (No Intervention): Subjects in the control group will be assessed in the same way and same time as the intervention group.

INTERVENTIONS:
Dietary Supplement: E+ — 300 ml E+ per day (525 kcal, 22.5 gram protein) for 35 days.
  Arms: E+ drink, enriched with energy and nutrients.

SUMMARY:
Malnutrition increases the risk of complications and predisposes ti infections through impaired immune response and wound healing. Healthcare costs related to the management of malnourished patients is estimated to be more than double the amount spent managing non- malnourished

The objective of this study is to examine the effect of newly developed energy and nutrients-dense beverage product on the nutritional status among patients at risk of malnutrition.

DETAILED DESCRIPTION:
Malnutrition is a complex state described as a deficiency of energy, protein and other nutrients causing measurable adverse effect on body tissue, function and clinical outcome.

Oral nutritional supplementation has in multiple individual trials and meta-analyzes shown an increased total energy intake and protein intake in patients in hospital settings as well as in the community.

The largest producer of dairy products in Norway, TINE AS released a new milk based energy- and nutrient dense product, called E+. The initiative behind this was Haukeland University Hospital and the municipality of Bergen. The product were developed to prevent malnutrition in the elderly and patients with a low food intake and high energy requirements.

The overall contribution to this study will be to provide new insight on how to offer malnourished patients the best available treatment.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of homecare services in the municipality of Bergen
* Recipients determined as at-risk of malnutrition based on screening with MNA (mini-nutritional assessment)
* Informed consent by participant
* Informed consent by participants and close relatives or guardian in case of dementia

Exclusion Criteria:

* Terminal care patients with < 3 month life expectancy
* Patients using parenteral or enteral nutrition
* Patients prescribed oral nutritional supplementation before recruitment
* Pregnancy
* Diabetes Mellitus
* Lactose intolerance
* Patients without a norwegian personal identification number
* Psychiatric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in Hand grip strength | Assessment at day 0, 35 and 70.
  Hand grip strength will be measured in kg with a handgrip dynamometer. Subjects will be asked to perform a maximal contraction for a few seconds with the non-dominant hand three times with about 10-20 seconds between each trial.
Change in Body weight | At day 0, 35 and 70
  Participants will be asked to remove shoes, socks, heavy clothing and jewelry for measurement of body weight to the nearest 100 g using portable digital scales.
Change in Body composition | At day 0, 35 and 70
  A Bioelectric impedance analysis will be used to calculate change in body composition. Measurements will be conducted by a device sending weak electric signals through the participant's body. The method is non-invasive and is commonly used by medical, health and fitness professionals.

SECONDARY OUTCOMES:
Change in Nutritional intake | At day 0, 35 and 70
  Dietary intake will be assessed for each study participant using a twenty-four-hour recall method conducted by the investigator and two additional people employed to help with the data collection. All three data collectors will use a standardized interview. The data collected will be used to calculate daily calorie and protein intake by entering the food records into a computerized version of a food composition table, Dietist XP.
Change in Quality of life | At day 0, 35 and 70
  Measurements of global subjective well-being and quality of life will be assessed using a simple visual analogue scale (VAS QL).

CONTACTS AND LOCATIONS:
Overall Officials: Randi J Tangvik, PhD-student, Study Chair — Clinical Dietitian at Haukeland University Hospital
Locations (1):
- Home Care Services, Bergen, Norway